CLINICAL TRIAL: NCT06719609
Title: Enovis High Ankle Sprain Brace Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Enovis Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-1684; Protocol Version 5/27/2025 (Other: UW Madison); A536130 (Other: UW Madison)
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-05

CONDITIONS: Athletes in Cutting Sports
Keywords: syndesmosis; ankle sprain; ankle bracing
MeSH Terms: conditions — Ankle Injuries | interventions — Hyaluronan Synthases; Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Running activity (Experimental): Participants will run for 1 minute at varying speeds
  Interventions: Other: Ankle tape; Other: Standard lace-up ankle brace; Other: Standard high ankle-sprain (HAS) brace; Other: Low-profile HAS brace; Other: No ankle brace or tape
- Dynamic agility task (Experimental): Participants will complete a 20-yard shuttle test
  Interventions: Other: Ankle tape; Other: Standard lace-up ankle brace; Other: Standard high ankle-sprain (HAS) brace; Other: Low-profile HAS brace; Other: No ankle brace or tape

INTERVENTIONS:
Other: Ankle tape — The influence of ankle tape on gait biomechanics
Other: Standard lace-up ankle brace — The influence of lace-up ankle brace on gait biomechanics
Other: Standard high ankle-sprain (HAS) brace — The influence of standard HAS brace on gait biomechanics
Other: Low-profile HAS brace — The influence of low-profile HAS brace on gait biomechanics
Other: No ankle brace or tape — The influence of no ankle tape or brace on gait biomechanics

SUMMARY:
The goal of this clinical trial is to learn if a new ankle brace impacts athletic motions. The main questions it aims to answer are:

* Does it impact motions such as running and cutting?
* Is it comfortable?

Researchers will compare 5 ankle bracing conditions.

Participants will:

* Perform a running activity
* Perform a cutting activity
* Complete a survey

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 at the time of data collection
* English-speaking
* Not currently pregnant
* No history of lower extremity surgery or chronic ankle instability
* No ankle injuries that required medical attention or ≥ 7 days of modified physical activity within the last 3 months
* Currently cleared for all physical activity
* Comfortable running on a treadmill for 10 minutes at a self-selected pace
* Have prior experience wearing an ankle brace and / or ankle tape during sport activities
* Shoe size US Men's 7.5-11.5 or Women's 9-13

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Comfort of bracing condition - treadmill activity | 90 minutes
  Participants will rate the comfort of each bracing condition. The comfort scale ranges from completely uncomfortable to completely comfortable.
Movement ability - treadmill activity | 90 minutes
  Participants will rate how each bracing condition impacted their ability to move. Movement scale ranges from no impact to completely changed my movement.
Ankle stability - treadmill activity | 90 minutes
  Participants will rate how stable their ankle felt in each bracing condition. Stability scale ranges from very stable to completely unstable.
Likelihood of use during sport - treadmill activity | 90 minutes
  Participants will rate how likely they are to use each bracing condition during their sport. Likelihood scale ranges from extremely unlikely to extremely likely.
Comfort of bracing condition - shuttle test | 90 minutes
  Participants will rate the comfort of each bracing condition. The comfort scale ranges from completely uncomfortable to completely comfortable.
Movement ability - shuttle test | 90 minutes
  Participants will rate how each bracing condition impacted their ability to move. Movement scale ranges from no impact to completely changed my movement.
Ankle stability - shuttle test | 90 minutes
  Participants will rate how stable their ankle felt in each bracing condition. Stability scale ranges from very stable to completely unstable.
Likelihood of use during sport - shuttle test | 90 minutes
  Participants will rate how likely they are to use each bracing condition during their sport. Likelihood scale ranges from extremely unlikely to extremely likely.
Ankle joint stability | 10 minutes
  Ultrasound will be used during Reverse Anterolateral Drawer Test. The examiner will hold the participant's foot stable against the exam table and will use their other hand to translate the participant's tibia/shank posteriorly. A second examiner will record an US video of the ankle joint during this test to measure the relative translation between the talus and the fibula. These procedures will be repeated on the other limb.

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Joachim, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes